CLINICAL TRIAL: NCT05557305
Title: Evaluation of the Usability, Safety, and Possible Beneficial Effects on Motor and Cognitive Functions Associated With Using a Neuro-rehabilitation Platform With Video Games in Pediatric Patients With Unilateral Spastic Cerebral Palsy
Brief Title: Changes in Motor and Cognitive Function on Unilateral Spastic Cerebral Palsy, Associated With Videogame Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: National Institute of Pediatrics, Mexico (Other Government)
Responsible Party: Principal Investigator, Ana María Escalante Gonzalbo, Head of the Laboratory of neurorehabilitation (LANR) IFC, UNAM, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/054
Record Dates: First submitted 2022-09-21; First posted 2022-09-28 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy, Spastic; Hemiplegia, Spastic
Keywords: virtual rehabilitation; video games; motor function; spastic hemiparesis; cerebral palsy; unilateral spastic cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia | interventions — Telerehabilitation; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Pilot, randomized, controlled, longitudinal trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videogame therapy (Experimental): The participants of the experimental group will only undergo video game therapy and will be called twice a week to perform supervised video game rehabilitation therapy, for a period of 45-50 minutes per session, for 10 weeks
  Interventions: Device: Videogame therapy
- Conventional therapy (Active Comparator): The participants in the control group will undergo the conventional therapy prescribed by their treating physician, at the INP they are prescribed occupational therapy, which is usually focused on game activities with balls, dice, cubes, tying ropes, etc., twice a week for 10 weeks.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Device: Videogame therapy — There will be 5 video game-type applications for virtual therapy, each with a specific therapeutic objective, which will be administered by trained personnel, depending on the characteristics of each patient.
  Other Names: Virtual rehabilitation
  Arms: Videogame therapy
Other: Conventional therapy — Occupational therapy with different play materials
  Other Names: Occupational therapy
  Arms: Conventional therapy

SUMMARY:
The use of interactive applications associated with position and movement sensors has begun to spread as an option for the reinforcement of physical rehabilitation therapies in patients with congenital or acquired motor disorders as a result of some neurological damage, due to its portability and the relative autonomy granted to the patient. However, the results of its effectiveness and impact continue to be scarce compared to the traditional therapy used for rehabilitation. The aim of this study is to explore possible benefits associated with occupational therapy with video games in patients with unilateral spastic cerebral palsy, comparing them with conventional therapy.

A randomized pilot study will be carried out, with a control group. The intervention will consist of the application of a virtual rehabilitation program for the experimental group while the control group will receive only conventional therapy. Before and after the said intervention, standardized tests will be applied to evaluate both motor function and the cognitive performance of the participants.

DETAILED DESCRIPTION:
This intervention protocol aims to validate five interactive applications for neurorehabilitation, as an effective therapeutic complement for the rehabilitation of children with unilateral cerebral palsy, compared to conventional rehabilitation.

The intervention contemplates first a phase of application of standardized tests in the Cognitive enablement lab of the National Institute of pediatrics (INP) in Mexico City, to determine, among other things, if the patient meets the established inclusion criteria. Patients who meet these criteria will be randomly assigned to the control or experimental group.

In the same INP, standardized tests will be applied to record their motor and cognitive capacity at the beginning of the protocol. Patients in the experimental group will receive two 50-minute video game rehabilitation sessions per week, for 10 weeks, under the supervision of trained personnel from the Laboratory of Applications for Neurorehabilitation (LANR). Control group patients will receive 10 weeks of occupational therapy, as prescribed by their treating physician.

All standardized tests will be applied again to the participants of both groups after the 10 weeks of intervention, and again six months later, to measure the persistence of the changes.

In the case of the experimental group, five interactive applications will be tested, each with a different sensor and virtual environment, as well as its own therapeutic objective, these applications are part of the National Autonomous University of Mexico (UNAM) virtual rehabilitation platform.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Both genders
* Reside in Mexico City and the metropolitan area
* Between 5 and 18 years old
* With upper extremity hemiparesis caused by Unilateral Spastic Cerebral Palsy (USCP) on their dominant side or not
* Who are at levels I-III of the Manual Ability Classification System for Children with Cerebral Palsy (MACS)
* Score equal to or greater than 20 on the Fugl-Meyer upper extremity scale.

Exclusion Criteria:

* Patients with joint instability (shoulder, elbow, or wrist)
* With severe concomitant medical problems such as congestive heart failure or seizures that prevent adequate attention to the task.
* Severe aphasia
* Hemineglect
* Visual disturbances that are not corrected with glasses
* Uncompensated hearing impairment
* Inability to understand instructions (Token Test < 17)
* Patients receiving concurrent therapies.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Fugl-Meyer Assesment for upper extremity (FMUE) | Baseline, 10 Weeks, 6 months
  Level of motor deficit, evaluated using the Fugl-Meyer Assessment scale for the upper limb (0-66), with 66 meaning no defficit.
Change in the Quality of Upper Extremity Skills Test (QUEST) | Baseline, 10 Weeks, 6 months
  Upper limb motor skill level, obtained through the Quality of Upper Extremity Skills Test (less than 0 to 100), with 100 being the best quality of movement.

SECONDARY OUTCOMES:
Change in the PedsQl pediatric quality of life questionnaire | Baseline, 10 Weeks, 6 months
  Level of independence in performing activities of daily living (ADLs), assessed using the PedsQl pediatric quality of life questionnaire (0-132) with 0 as the highest score.
Change in the digital version of the Trail Making Test (TMT-A) | Baseline, 10 Weeks, 6 months
  Changes in cognitive function in terms of speed of executive functions and attention, measured by a digitized version of the Trail Making Test A.
Change in the digital version of the Corsi cube test. | Baseline, 10 Weeks, 6 months
  Changes in working memory measured by the Corsi Cubes test.
Change in the digital version of the Perception of differences test (FACES) | Baseline, 10 Weeks, 6 months
  Changes in visual perception, using the perception of differences test
Change in the Digital implementation of the Go-NoGo paradigm. | Baseline, 10 Weeks, 6 months
  Changes in inhibition and flexibility functions, measured using a digital implementation of the Go-NoGo paradigm

CONTACTS AND LOCATIONS:
Overall Officials: Ana María Escalante-Gonzalbo, MCompSci, Principal Investigator — National University of Mexico
Locations (1):
- Instituto Nacional de Pediatría, Mexico City, Coyoacán, CDMX, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Escalante-Gonzalbo AM, Ramirez-Graullera YS, Pasantes H, Aguilar-Chale JJ, Sanchez-Castillo GI, Escutia-Macedo XA, Briseno-Soriano TM, Franco-Castro P, Estrada-Rosales AL, Vazquez-Abundes SE, Andrade-Morales D, Hernandez-Franco J, Palafox L. Safety, Feasibility, and Acceptability of a New Virtual Rehabilitation Platform: A Supervised Pilot Study. Rehabil Process Outcome. 2021 Aug 7;10:11795727211033279. doi: 10.1177/11795727211033279. eCollection 2021. PMID 34987304
- See also: Web Page of the Research and Development Laboratory of Interactive Applications for Neuro-Rehabilitation (LANR) of the UNAM — http://lanr.ifc.unam.mx